CLINICAL TRIAL: NCT07224022
Title: NACho: A Study of Neo-Adjuvant Cemiplimab With Fianlimab for Resectable Non-Metastatic Colon Cancer
Brief Title: Cemiplimab With Fianlimab for Resectable Non-Metastatic Colon Cancer
Acronym: NACho
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: John Strickler, M.D. (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, John Strickler, M.D., Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00118775
Record Dates: First submitted 2025-10-30; First posted 2025-11-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Colon Cancer
Keywords: Previously untreated; pMMR; MSS; Neoadjuvant; Resectable; Non-metastatic; previously untreated T4N0 or stage III pMMR/MSS colon cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — cemiplimab

STUDY DESIGN:
Intervention Model Description: The study will be conducted in two stages: 1) Safety Run-In Cohort; 2) Expansion Cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cemiplimab in combination with Fianlimab (Experimental): All patients will be treated with fianlimab 1600 mg IV plus cemiplimab 350 mg IV on Days 1 and 22.
  Interventions: Drug: Cemiplimab + Fianlimab [Fixed Dose Combination (FDC)]

INTERVENTIONS:
Drug: Cemiplimab + Fianlimab [Fixed Dose Combination (FDC)] — Immune checkpoint inhibition with antibodies directed against PD-1 and CTLA-4 receptors have demonstrated significant and durable efficacy in several advanced malignancies. LAG-3 is classified as an immune checkpoint protein that negatively regulates T cell activity, similar to PD-1 and CTLA-4. Blockade of LAG-3 with antibodies such as fianlimab, especially in combination with anti-PD-1 therapy, may represent a potentially effective or enhanced treatment for advanced malignancies.
  We hypothesize that cemiplimab in combination with fianlimab is feasible, safe, and effective neoadjuvant treatment strategy for early-stage colon cancer.

SUMMARY:
This is a research study to test whether two immunotherapy drugs-cemiplimab and fianlimab-can safely and effectively shrink colon tumors before surgery in people with stage II-III colon cancer that has not spread to other parts of the body.

Participants will receive two doses of the study drugs through an IV (one on Day 1 and one on Day 22). During the study, participants will have regular visits to the study clinic and multiple tests for safety and research purposes, including blood tests, along with other tests and scans, followed by surgery to remove the tumor. The study will follow participants' health for up to three years after surgery.

Risks of cemiplimab and fianlimab include fatigue, diarrhea, skin rash, thyroid problems, and immune-related side effects such as inflammation of the lungs, liver, or intestines.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, phase II study to assess the safety, feasibility, and clinical activity of cemiplimab with fianlimab in patients with resectable colon cancer. All patients will be treated with fianlimab 1600 mg IV plus cemiplimab 350 mg IV on Days 1 and 22. The study will be conducted in two stages: 1) Safety Run-In and 2) Expansion. Approximately 24 patients will be enrolled to ensure 20 evaluable patients.

All patients will complete a medical history, baseline physical examination, and clinical assessment including laboratory studies prior to starting treatment. Physical examination, evaluation of AEs, and safety labs will be conducted while on treatment. Toxicities will be recorded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 6.0. All study assessments will be conducted as per the study calendar.

All patients will undergo baseline tumor staging consisting of imaging of the chest, abdomen, and pelvis. Pretreatment tumor biopsies will be taken during colonoscopies. All patients should receive surgical resection of the colon primary from 30 to 60 days after Day 1, unless medically contraindicated or the patient withdraws/is withdrawn from study. Post-treatment tissue is obtained at surgery. Patients may receive adjuvant chemotherapy as per standard of care. Adjuvant chemotherapy may be considered for patients with pathologic stage II/III disease approximately 6-12 weeks after surgery unless medically contraindicated or the patient withdraws/is withdrawn from study. Patients will be followed for recurrence and survival for up to 3 years. Recurrence will be determined by medical provider assessment. Survivorship will be followed according to national guidelines and institutional standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and/or cytologically documented adenocarcinoma of the colon
2. Tumor testing indicating proficient mismatch repair and/or microsatellite stable (pMMR/MSS)
3. No evidence of measurable distant metastatic disease (as per RECIST v1.1 criteria) based on CT of the chest, abdomen, and pelvis
4. T4N0 or stage III colon cancer as per baseline CT imaging (see Appendix E for imaging guidelines)
5. Candidate for surgical resection with curative intent
6. Age ≥ 18 years
7. ECOG Performance Score of 0 or 1
8. Adequate marrow function as evidenced by:

   1. Absolute neutrophil count (ANC) ≥ 1,500/µL
   2. Platelets ≥ 100,000/µL
   3. Hemoglobin (Hgb) ≥ 8 g/dL
9. Adequate renal function as evidenced by either calculated CrCL ≥ 50 mL/min using the Cockcroft-Gault formula or serum creatinine <1.5x upper limit of normal (ULN)
10. Adequate hepatic function as evidenced by:

    1. Total serum bilirubin < 1.5 x ULN unless conjugated bilirubin ≤ ULN (conjugated bilirubin only needs to be tested if total bilirubin exceeds ULN)
    2. Aspartate aminotransferase (AST) ≤ 2.5 x ULN
    3. Alanine aminotransferase (ALT) ≤ 2.5 x ULN
    4. Alkaline phosphatase ≤ 3 x ULN
11. Ability to undergo colonoscopy with biopsies after registration to obtain study-specific tissue. Note: If colonoscopy and/or biopsies are not possible, the subject will be excluded.
12. Women of childbearing potential (WOCBP) must have a negative serum (beta-hCG) at screening.

    1. WOCBP are defined as women who are fertile following menarche until becoming postmenopausal, unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy.

       A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high FSH level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient to determine the occurrence of a postmenopausal state. The above definitions are according to the CTFG guidance. Pregnancy testing and contraception are not required for women with documented hysterectomy.
    2. Male study participants with WOCBP partners are required to use condoms during the study and until 6 months after the last dose of study treatment unless they are vasectomized or practice sexual abstinence.
    3. Vasectomized partner or vasectomized study participant must have received medical assessment of the surgical success.
    4. Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and LAM are not acceptable methods of contraception. Female condom and male condom should not be used together.
13. WOCBP must agree not to donate eggs (ova, oocytes) for the purpose of assisted reproduction during the entire trial and until 6 months after last treatment
14. All men must agree not to donate sperm during the trial and for 6 months after receiving the last therapy dose
15. Patients or their legal representatives must be able to read, understand and provide informed consent to participate in the trial.

Exclusion Criteria:

1. Any previous treatment with immune checkpoint inhibitors targeting CTLA-4, PD-1 or PD-L1, or LAG3.
2. Any previous surgery, chemotherapy, radiotherapy or targeted therapy for colon or rectal cancer.
3. Clinical or radiographic evidence of bowel obstruction or perforation.
4. In the opinion of the Principal Investigator, any medical condition (e.g., significant gastrointestinal bleeding, symptomatic disease) that would preclude participation in study activities (e.g., colonoscopy, immunotherapy, surgery).
5. Uncontrolled pain related to primary colon malignancy.
6. Radiotherapy to the primary tumor prior to or planned post-surgery.
7. Gastrointestinal bleeding requiring a blood transfusion within 30 days of screening.
8. Treatment with another investigational device or study drug or participation in another drug study within 30 days of screening. Other investigational procedures while participating in this study are excluded.
9. Known hypersensitivity to the active substances or to any of the excipients.
10. History of myocarditis.
11. Troponin I TnI >2x institutional ULN at baseline. Patients with TnI levels between >1 to 2x ULN are permitted if repeat levels within 24 hours are ≤1x ULN. If TnI levels are >1 to 2x ULN within 24 hours, the subject may undergo a cardiac evaluation and may be considered for treatment by the investigator based on the medical judgement in the patient's best interest.
12. Intercurrent illnesses, including but not limited to active infections, unstable angina pectoris, symptomatic cardiovascular disease, or symptomatic congestive heart failure.
13. Uncontrolled infection, including HIV, HBV, or HCV; or diagnosis of immunodeficiency that is related to or results in chronic infection.

    1. Patients with known HIV who have controlled infection (undetectable viral load and CD4 count above 350 either spontaneously or on a stable antiviral regimen) are permitted. For patients with controlled HIV infection, monitoring will be performed per local standards.
    2. Patients with known hepatitis B (HepBsAg+) who have controlled infection (serum hepatitis B virus DNA PCR that is below the limit of detection AND receiving anti-viral therapy for hepatitis B) are permitted. Patients with controlled infections must undergo periodic monitoring of HBV DNA per local standards and must remain on anti-viral therapy for at least 6 months beyond the last dose of investigational study drug.
    3. Patients who are known hepatitis C virus antibody positive (HCV Ab+) who have controlled infection (undetectable HCV RNA by PCR either spontaneously or in response to a successful prior course of anti-HCV therapy) are permitted.
    4. Patients with HIV or hepatitis must be reviewed by a qualified specialist (e.g., infectious disease or hepatologist) managing this disease prior to and regularly throughout the duration of their participation in the trial
14. History of Crohn's disease, ulcerative colitis, or inflammatory bowel disease.
15. Ongoing or recent (within 2 years) evidence of an autoimmune disease that required systemic treatment with immunosuppressive agents. The following are non-exclusionary: vitiligo, childhood asthma that has resolved, residual hypothyroidism that requires only hormone replacement, psoriasis not requiring systemic treatment.
16. Is on chronic systemic steroids (>10 mg/day of prednisone or equivalent).

    1. Physiologic corticosteroid replacement therapy at doses >10 mg/day of prednisone or equivalent for adrenal or pituitary insufficiency and in the absence of active autoimmune disease is permitted.
    2. Participants with a condition (e.g., asthma or COPD) that requires intermittent use of bronchodilators, inhaled corticosteroids, or local corticosteroid injections may participate.
    3. Participants using topical, ocular, intra-articular, or intranasal corticosteroids (with minimal systemic absorption) may participate.
    4. Brief courses of corticosteroids for prophylaxis (e.g., contrast dye allergy) or study treatment-related standard premedications are permitted.
17. History of allogeneic organ transplant, including allogeneic stem cell transplantation.
18. Received a live vaccine within 30 days of planned start of study medication. If a patient intends to receive a COVID-19 vaccine before the start of study drug, participation in the study should be delayed at least 1 week after any COVID-19 vaccination. During the treatment period, it is recommended to delay COVID-19 vaccination until patients are receiving and tolerating a steady dose of study drug. A vaccine dose should not be less than 48 hours before or after study drug dosing.
19. History or current evidence of significant (CTCAE grade ≥2) local or systemic infection (e.g., cellulitis, pneumonia, septicemia) requiring systemic antibiotic treatment within two weeks prior to the first dose of trial medication.
20. Subjects with any previously untreated or concurrent cancer that is distinct in primary site or histology from colon except treated cervical cancer in-situ, treated non-metastatic skin cancer, treated prostate cancer, or treated superficial bladder tumor.

    Note: Subjects surviving a cancer that was curatively treated and without evidence of disease or biochemical relapse (undetectable PSA for prostate cancer) for 2 or more years before registration are allowed. All cancer treatments must be completed at least 2 years prior to registration.
21. Female subjects who are pregnant or breast-feeding, or planning to become pregnant during study treatment or through 6 months after dose of study drugs.
22. Women of childbearing potential (WOCBP) who are unwilling to practice highly effective contraception prior to the initial dose/start of the first treatment, during the study, and for at least 6 months after the last dose. Highly effective contraceptive measures include:

    1. Stable use of combined (estrogen and progestogen containing) hormonal contraception (oral, intravaginal, transdermal) or progestogen-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation initiated 2 or more menstrual cycles prior to screening;
    2. Intrauterine device; intrauterine hormone-releasing system;
    3. Bilateral tubal occlusion/ ligation;
    4. Vasectomized partner (provided that the male vasectomized partner is the sole sexual partner of the WOCBP study participant and that the vasectomized partner has obtained medical assessment of surgical success for the procedure); and/or
    5. Sexual abstinence†, ‡. Pregnancy testing and contraception are required for WOCBP. Pregnancy testing and contraception are not required for women who are post-menopausal or permanently sterile.

    A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high FSH level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient to determine the occurrence of a postmenopausal state. The above definitions are according to the CTFG guidance.

    †Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study drugs. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject.

    ‡Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and LAM are not acceptable methods of contraception. Female condom and male condom should not be used together.
23. Evidence of interstitial lung disease, history of interstitial lung disease, or active, noninfectious pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility of treatment with cemiplimab and fianlimab before surgery | 60 days after first study treatment
  Measured by the proportion of patients completing surgery within 60 days after Day 1 of treatment with cemiplimab and fianlimab
Safety of treatment with cemiplimab and fianlimab before surgery | AEs will be assessed from Day 1 through Day 112 (90 days after the last dose of study treatment)
  The frequency and severity of adverse events, according to NCI CTCAE V6.0

SECONDARY OUTCOMES:
Two-year disease-free survival | Up to two years after surgery
  Measured from surgery until documented disease recurrence among patients with R0 resection and no known metastatic disease following resection of the primary tumor
Pathological Response | Resection is to occur from 30 to 60 days after the first dose of study drug
  Measurement of residual viable tumor at the time of resection

IPD SHARING:
Plan to Share IPD: No